CLINICAL TRIAL: NCT04285970
Title: Analysis of the Motion Activity Manual Wheelchair Users
Acronym: Acti-FRM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190373
Record Dates: First submitted 2020-02-17; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2019-07

CONDITIONS: Spinal Cord Injuries
Keywords: detection rate of propulsion cycles
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medullary injured: Injured Medullary users of manually driven wheelchairs for daily locomotion
  Interventions: Other: detection of effort intensity
- Healthy volunteers: Healthy volunteer with at least 2 hours' experience using a manual wheelchair
  Interventions: Other: cycle detection

INTERVENTIONS:
Other: cycle detection — 6-minute test on a treadmill at pedestrian speed (5km/h) with 2 instruments (dynamometric wheel and inertial centre) on a standardised wheelchair
  Groups: Healthy volunteers
Other: detection of effort intensity — 6-minute test on an urban course with 2 instruments (dynamometric wheel and inertial units) on a wheelchair
  Groups: Medullary injured

SUMMARY:
Currently, there is no system in place to allow manual wheelchair users to know their quantities of movement activities and the intensity of effort to be provided during these propulsion movements. Based on recent work by Routhier et al. in 2017, and in light of the scientific literature related to wheelchair propulsion, it would seem appropriate to validate the use of inertial units as tools to quantify and categorize the intensity of manual wheelchair propulsion.

DETAILED DESCRIPTION:
The investigator hypothesize that an inertial unit positioned on the wheelchair wheel has the same detection rate of the propulsion cycle as a dynamometric wheel (step 1). In addition, the investigator hypothesize that the categorization of the detected propulsion cycle as a function of force intensity is similar between the angular deceleration of the wheel during propulsion calculated from the inertial unit and the external mechanical power calculated from a dynamometric wheel (step 2).

ELIGIBILITY:
Inclusion Criteria:

For the healthy user group volunteers:

* Men or women over 18 years of age,
* An experience of at least 2 hours using the manual wheelchair,
* Subject who has signed an informed and written consent,
* Affiliation to a social security system.

For the spinal cord injured user group:

* Men or women over 18 years of age,
* Injured Medullary users of manually propelled wheelchairs for daily locomotion (at least 30/100 at WST on travel items),
* Subject who has signed an informed and written consent,
* Affiliation to a social security system.

Exclusion Criteria:

* Patient refusing to participate in the study,
* Manual wheelchair users with propulsion assistance system,
* Major cognitive disorders,
* Unbalanced cardiovascular disease,
* Pressure sores and unhealed palm lesions,
* Asthma to effort,
* Progressive etiologies: tumor, infectious, inflammatory and associated - - pathologies: head trauma, amputation,
* Patient under guardianship or curatorship,
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Manuel wheelchair users
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Confirm the identification of propulsion cycles during a journey at constant speed (5km/h) | 18 months
  Measurement of the detection rate of propulsion cycles
Confirm the classification of propulsion cycles by effort intensity | 18 months
  Classification rate of propulsion cycles

SECONDARY OUTCOMES:
Study of the association between the propulsion force and the coefficient of the deceleration slope | 18 months
  The association will be measured with propulsion force by the torque wheel and the coefficient of the deceleration slope quantified by the inertial unit

CONTACTS AND LOCATIONS:
Overall Officials: URC PIFO, Study Director — Assistance Public - Hôpitaux de Paris
Locations (1):
- Raymond Poincaré Hospital - Spinal Cord Injury Unit, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boninger ML, Cooper RA, Baldwin MA, Shimada SD, Koontz A. Wheelchair pushrim kinetics: body weight and median nerve function. Arch Phys Med Rehabil. 1999 Aug;80(8):910-5. doi: 10.1016/s0003-9993(99)90082-5. PMID 10453767
- [Background] Boninger ML, Souza AL, Cooper RA, Fitzgerald SG, Koontz AM, Fay BT. Propulsion patterns and pushrim biomechanics in manual wheelchair propulsion. Arch Phys Med Rehabil. 2002 May;83(5):718-23. doi: 10.1053/apmr.2002.32455. PMID 11994814